CLINICAL TRIAL: NCT03532607
Title: The Impact of Music Meditation Therapy on Pain, Mood, and Stress When Botulium Toxin (Botox) Injection is Utilized: A Randomized Controlled Trial
Brief Title: The Effect of Music Meditation Therapy in Patients With Chronic Pain Receiving Botox
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rowan University (Other)
Responsible Party: Principal Investigator, Richard Jermyn, Director, NeuroMusculoskeletal Institute, Rowan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro2015000590
Record Dates: First submitted 2015-12-21; First posted 2018-05-22 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Pain
Keywords: Chronic
MeSH Terms: conditions — Pain; Bronchiolitis Obliterans Syndrome | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Participants will be asked to listen to pre-recorded music offered by the research team from an ipod for 30 minutes. After the 30 minutes have elapsed, the research staff will return and ask the patient to turn off the music. The patient then will be escorted to the clinic room to receive the botox injection.
  Interventions: Other: Music
- Control (No Intervention): After completing the consent form, the participants who are assigned to the control group will be asked to remain in the patient waiting area. The patient then will be escorted to the clinic room to receive the botox injection.

INTERVENTIONS:
Other: Music — Patients will listen to soothing music for 30 minutes before their standard of care botox injection
  Arms: Treatment

SUMMARY:
The purpose of this pilot study is to examine the impact of music meditation therapy session on patients with chronic pain who are receiving Botox injections at a pain management center.

DETAILED DESCRIPTION:
This study is a randomized controlled trial (RCT) that employs a two-arm parallel-group design. Ninety-eight participants scheduled to receive a Botox injection will be randomly assigned to receive individual music meditation therapy intervention group or standard care control group before the participant's Botox injection. The study team will use an embedded mixed methods study that uses both quantitative and qualitative data. Qualitative data play a supporting role and are embedded within a larger RCT. The qualitative data will help the investigators better understand the patients' experience of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both genders ages 18-60 who have been referred for Botox injection for treatment of chronic pain at the Rowan SOM NeuroMusculoskeletal Institute. These patients will have a prior diagnosis made by their physicians necessitating treatment with Botox injections.
* Patients who have previously received a Botox injection or patients receiving Botox injections for the first time can participate.

Exclusion Criteria:

* Patients who cannot speak or understand English for informed consent and patient teaching
* Patients with hearing impairment.
* Pregnant women, children and/or minors, cognitively impaired patients or the elderly (above 60 years of age).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2015-12; Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Pain Visual Analogue Scale (VAS) | 3 minutes
  The VAS is a 100-mm line, the length of which represents a continuum of an experience such as pain. Verbal descriptors mark the end of the continuum. The study team use the verbal descriptors 'no pain' and 'worst imaginable pain.'

SECONDARY OUTCOMES:
Stress Visual Analogue Scale (VAS) | 3 minutes
  The VAS is a 100-mm line, the length of which represents a continuum of an experience such as stress. Verbal descriptors mark the end of the continuum. The study team use the verbal descriptors 'no stress' and 'extreme stress.'
Mood Visual Analogue Scale (VAS) | 3 minutes
  The VAS is a 100-mm line, the length of which represents a continuum of an experience such as mood. Verbal descriptors mark the end of the continuum.The study team use the verbal descriptors 'best mood' and 'worst mood.'

CONTACTS AND LOCATIONS:
Overall Officials: Richard Jermyn, DO, Principal Investigator — Rowan University School of Osteopathic Medicine
Locations (1):
- Rowan University SOM NeuroMusculoskeletal Institute, Stratford, New Jersey, United States